CLINICAL TRIAL: NCT04641312
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3457263 in Healthy Participants and in Patients With Type 2 Diabetes
Brief Title: A Study of LY3457263 in Healthy Participants and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17261; 2020-001828-34 (EudraCT Number); J1R-MC-GZFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01-01

CONDITIONS: Healthy; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- LY3457263 - Part A (Experimental): Escalating single doses of LY3457263 administered subcutaneously (SC) to healthy participants
  Interventions: Drug: LY3457263
- Placebo - Part A (Placebo Comparator): Placebo administered SC to healthy participants
  Interventions: Drug: Placebo
- LY3457263 - Part B (Experimental): Escalating single doses of LY3457263 administered SC in combination with Dulaglutide administered SC to participants with type 2 diabetes
  Interventions: Drug: LY3457263; Drug: Dulaglutide
- Placebo - Part B (Placebo Comparator): Placebo administered SC in combination with Dulaglutide administered SC to participants with type 2 diabetes
  Interventions: Drug: Dulaglutide; Drug: Placebo

INTERVENTIONS:
Drug: LY3457263 — Administered SC
  Arms: LY3457263 - Part A; LY3457263 - Part B
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: LY3457263 - Part B; Placebo - Part B
Drug: Placebo — Administered SC
  Arms: Placebo - Part A; Placebo - Part B

SUMMARY:
The main purpose of this study is to investigate the safety and tolerability of the study drug LY3457263 in healthy participants and participants with type 2 diabetes. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. The study has two parts (part A and B). Each part will last up to 10 weeks and may include up to either 13 (part A) or 19 (part B) visits.

ELIGIBILITY:
Inclusion Criteria:

* Males that agree to use an effective method of contraception or agree to remain abstinent
* Females that are not of childbearing potential due to postmenopausal status or due to surgical sterility
* Part A only:

  * Are overtly healthy
  * Body mass index (BMI) of 18.5 to 35 kilograms per meter squared (kg/m²)
* Part B only:

  * Have been diagnosed with Type 2 Diabetes (T2D) for at least 6 months prior to screening
  * Be treated for T2D with stable dose of metformin, a stable dose of a dipeptidyl peptidase-4 (DPP-4) inhibitor with or without metformin, or a stable dose of a glucagon-like peptide-1 (GLP-1) receptor agonist with or without metformin for at least 3 months prior to screening
  * BMI of 27 to 40 kg/m²

Exclusion Criteria:

* Have undergone any form of bariatric surgery

  * Have used or intend to use medications that promote weight loss within 3 months prior to screening, for the duration of the study
  * Part A only:

    * Have fasting plasma glucose (PG) levels ≥7 millimoles per liter (mmol/L) (≥126 milligrams per deciliter (mg/dL)) at screening
    * Have Hemoglobin A1c (HbA1c) level ≥ 6.5% (48 millimoles per mole (mmol/mol)) at screening
    * Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >20% and 10%, above the upper limit of normal (ULN), respectively. Elevation of total bilirubin level is considered acceptable in case of Gilbert's disease (with a normal direct bilirubin)
  * Part B only:

    * Have Type 1 Diabetes or latent autoimmune diabetes in adults
    * Have uncontrolled diabetes defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization in the 6 months prior to screening
    * Have known proliferative diabetic retinopathy, diabetic maculopathy, or severe nonproliferative diabetic retinopathy
    * Present comorbid conditions commonly associated with diabetes (for example, hypertension, hypercholesterolemia, hypothyroidism) unless they are well-controlled with stable medication
    * Have had an episode of severe hypoglycaemia within 6 months prior to screening, or have a history of hypoglycaemia unawareness or poor recognition of hypoglycaemia
    * Have a history of acute or chronic pancreatitis or elevation in serum lipase and/or amylase >2 × ULN at screening
    * Have a resting heart rate of <50 or >100 beats per minute
    * Have an estimated glomerular filtration rate (<60 milliliter/minute (mL/min)/1.73 m2, or a level of estimated glomerular filtration rate that would contraindicate the use of metformin per the label in the respective country
    * Have a screening calcitonin ≥20.0 picograms per milliliter (pg/mL)
    * Fasting serum triglyceride level of >500 mg/dL at screening
    * Have serum AST or ALT >3 × ULN or TBL >1.5 × ULN (except for participants diagnosed with Gilbert's syndrome)
    * Have taken any prescription medication that are specifically indicated for lowering serum triglycerides within the last 3 months
    * Have taken within the last 3 months any medications that interfere with absorption of dietary cholesterol or fats
    * Use of medications known to prolong the QT/QTc interval
    * Treated only with diet and exercise at study entry

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 42
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3457263 | Day 1 through Day 42
  PK: AUC[0-inf] of LY3457263

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- Germany (2):
  - Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia
  - Profil Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No